CLINICAL TRIAL: NCT06673706
Title: Assessing the Impact of Front-of-package Nutrient Labels on Consumer Understanding and Behavior
Brief Title: Assessing the Impact of Front-of-package Nutrient Labels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Jennifer Falbe, Associate Professor, University of California, Davis
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 1641776-8B
Record Dates: First submitted 2024-10-24; First posted 2024-11-05 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Nutrition Knowledge; Attitudes; Dietary Habits; Dietary Behavior
MeSH Terms: conditions — Behavior; Feeding Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- No-label Control (No Intervention): Participants will see packaged food-and-beverage items with no front-of-package labels (other than any posted by the manufacturer).
- High-In with color (Experimental): Participants will see packaged food-and-beverage items displaying front-of-package labels that say, "High In [nutrient]" (nutrients: saturated fat, sodium, or added sugar) if the item contains 20% or more of the daily recommended limit per serving for each nutrient. The nutrients will be highlighted in red.
  If the item is not high in 1 or 2 of the nutrients, the nutrient(s) will not be on the label. If the item is not high in any of the 3 nutrients, the product will not display this label.
  Interventions: Other: Front-of-package label
- High-In black and white (Experimental): Participants will see packaged food-and-beverage items displaying front-of-package labels that say, "High In [nutrient]" (nutrients: saturated fat, sodium, or added sugar) if the item contains 20% or more of the daily recommended limit per serving for each nutrient. The label will have a white background and black text.
  If the item is not high in 1 or 2 of the nutrients, the nutrient(s) will not be on the label. If the item is not high in any of the 3 nutrients, the product will not display this label.
  Interventions: Other: Front-of-package label
- Nutrition Info with color (Experimental): Participants will see packaged food-and-beverage items displaying front-of-package labels that list "high", "medium", or "low" for saturated fat, sodium, and added sugars. "High" is defined as 20% or more of the daily recommended limit per serving, "medium" as 6-19%, and "low" as 5% or less. The word "high" will be highlighted red; the word "medium" will be highlighted yellow; and the word "low" will be highlighted green.
  Interventions: Other: Front-of-package label
- Nutrition Info black and white (Experimental): Participants will see packaged food-and-beverage items displaying front-of-package labels that list "high", "medium", or "low" for saturated fat, sodium, and added sugars. "High" is defined as 20% or more of the daily recommended limit per serving, "medium" as 6-19%, and "low" as 5% or less. The label will have a white background and black text.
  Interventions: Other: Front-of-package label
- Nutrition Info without color, with percent Daily Value (Experimental): Participants will see packaged food-and-beverage items displaying front-of-package labels that list "high", "medium", or "low" for saturated fat, sodium, and added sugars. "High" is defined as 20% or more of the daily recommended limit per serving, "medium" as 6-19%, and "low" as 5% or less. The label will also list the exact percent of the daily recommended limit (i.e., daily value) for each nutrient per serving. The label will have a white background and black text.
  Interventions: Other: Front-of-package label

INTERVENTIONS:
Other: Front-of-package label — Participants will see packaged food-and-beverage items displayed with labels as specified by their assigned group
  Arms: High-In black and white; High-In with color; Nutrition Info black and white; Nutrition Info with color; Nutrition Info without color, with percent Daily Value

SUMMARY:
This study aims to compare different front-of-package label designs, using two schemes: (1) High In and (2) Nutrition Info with each scheme having (1) a version with colors (i.e., green, yellow, and/or red) indicating level of nutrient content and (2) a black-and-white version. Additionally the Nutrition Info scheme will have a version that includes the percent Daily Value in black and white. Labels will be compared against a no-label control and one another.

DETAILED DESCRIPTION:
This study aims to compare different front-of-package label designs, using two schemes: (1) High In and (2) Nutrition Info. The labels will have variations, such as color, and will be compared to a no-label control and one another. There will be a total of 6 experimental conditions: 1) High In label with color; 2) High In label in black and white; 3) Nutrition Info label with color; 4) Nutrition Info in black and white; 5) Nutrition Info label in black and white with percent Daily Value listed; and 6) a no-label control.

Participants will view a series of food-and-beverage products labeled (or not) according to condition. The three primary outcomes are: (1) correct assessment of high nutrient contents in food-and-beverage products, (2) perceived healthfulness of packaged foods and beverages, and (3) selection of at least one item high in at least one nutrient of concern (saturated fat, sodium, added sugar) in a shopping task. Perceived message effectiveness will be examined as a secondary outcome.

All statistical analyses will use two-tailed tests with a significance level of <0.05. Per CONSORT Guidelines, all models comparing labels will be bivariate, regressing outcomes on indicators for labeling condition. For continuous outcomes, linear regression models will be used, and for dichotomous outcomes, risk ratios (or probability ratios) will be estimated using Poisson regression with a robust error variance.

Effect modification of the labels on primary outcomes will be explored for type 2 diabetes status and sociodemographic variables important for health equity using interaction terms and stratified models.

Additionally, differences in the primary outcomes between each of the 6 unique conditions will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Equal or greater than 18 years of age
* English-speaking
* U.S. residents
* Have eaten restaurant food at least once in the last month
* Participants will reflect the U.S. Census Bureau's 2021 American Community Survey 5-year estimates for gender, race/ethnicity, educational attainment, and age

Exclusion Criteria:

* Failing the attention check question
* Completing the survey in less than 33% of the median completion time

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10601 (Actual)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Correct assessment of "high" nutrients | Within approximately 5 minutes of intervention exposure
  Participants will view 4 foods and indicate whether each food is high in each of saturated fat, sodium, and added sugar. A "correct" response is identifying a high-in product as high in the corresponding nutrient and identifying a not high-in product as not high in the corresponding nutrient; otherwise the response is "incorrect". Participants will provide 12 responses (3 nutrients across 4 foods), and the percent correct for each participant will be used as a continuous outcome in linear regression. If the distribution of percent correct is skewed, analysis may use all 12 dichotomous responses in a mixed model, accounting for within subject correlation. In sensitivity analyses, this outcome will be (1) examined by nutrient and (2) dichotomized as correct assessment of all nutrients in each meal.
Perceived healthfulness | Within approximately 5 minutes of intervention exposure
  Participants will provide a healthfulness score (response scale from 1-7) for up to 6 different products. The average score across products will be used as a continuous outcome in linear regression models. In sensitivity analyses, scores will be examined by product and product grouping.
Selection of a product high in a nutrient of concern | Within approximately 5 minutes of intervention exposure
  Participants will select a food and beverage they would purchase for themselves from hypothetical grocery store shelves displaying foods and beverages. The dichotomous outcome is selection of an item that is high in at least one nutrient of concern (compared to not selecting an item high in at least one nutrient of concern), examined overall and separately for foods and beverages. Analyzed in Poisson regression with robust SE to directly estimate risk ratios.

SECONDARY OUTCOMES:
Perceived message effectiveness | Within approximately 5 minutes of intervention exposure
  Measured with one item from the validated 3-item University of North Carolina perceived message effectiveness scale: "How much does this label discourage you from wanting to consume products high in sodium, saturated fat, and added sugar?" Response options include 1-5 where higher values represent higher perceived discouragement. Analyzed as a continuous outcome in linear regression.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Falbe, ScD, MPH, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No